CLINICAL TRIAL: NCT02412553
Title: Dietary Therapy and Gut Microbiome in Crohn's Disease and Ulcerative Colitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ashwin Ananthakrishnan, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P001134
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Food, Formulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specific carbohydrate arm (Active Comparator): The specific carbohydrate diet will be sufficient to meet 100% of the caloric requirements of the patient.
  Interventions: Other: Specific carbohydrate diet
- Elemental diet arm (Active Comparator): The partial elemental diet will be sufficient to provide 50% of the daily caloric needs for each patient with the remainder from a standard low-residue diet
  Interventions: Other: Elemental diet

INTERVENTIONS:
Other: Specific carbohydrate diet
  Arms: Specific carbohydrate arm
Other: Elemental diet
  Arms: Elemental diet arm

SUMMARY:
The study is proposed as a 2-year single site, open-label clinical trial of enteral nutrition or the specific carbohydrate diet in patients with active CD or UC. Patients seeking care in the outpatient clinics of the Division of Gastroenterology at Massachusetts General Hospital will be approached for participation in the trial during their routine outpatient appointments. All patients are required to have a diagnosis of CD or UC confirmed using standard clinical, endoscopic, and histologic criteria. Eligible patients will complete an office visit to confirm eligibility for the study and informed consent will be obtained. They will then be scheduled for a routine colonoscopy as part of their standard clinical care to objectively confirm active disease and obtain biopsies for microbiome and gene expression. The investigators will obtain prior authorization from the subject's insurance company for such colonoscopy, or if it is not covered by the insurance, the investigators will use study funds to pay for the procedure. They will then be assigned to one of two dietary intervention arms based on their preference and will meet with the study registered dietician at the MGH Clinical Research Center (CRC) metabolism and nutrition unit. There, they will receive instruction on the components of the assigned dietary therapy arm - partial elemental diet (enteral nutrition) or specific carbohydrate diet, and will complete a baseline food record (FR). They will adhere to the dietary therapy for 6 weeks after which they can resume normal diet. Clinical, biochemical, nutritional, and microbiological parameters will be measured during and for 6 weeks following the study. They will have 5 study visits during this time.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Able to provide written informed consent prior to screening and to comply with the requirements of the study protocol.
3. Established diagnosis of small bowel or colonic CD or ulcerative colitis
4. Confirmation of active CD or UC with recent (within 1 month) objective evidence of active disease on colonoscopy
5. Any medications being currently used for IBD must remain stable during the study period with the exception of tapering of corticosteroids.
6. Current disease activity defined as a Harvey Bradshaw index > 4 at baseline (week 0) or SCCAI > 3

Exclusion Criteria:

1. If female, is pregnant or is breast feeding
2. Known celiac disease or subjects with a positive screen for celiac disease (elevated tissue transglutaminase antibodies)
3. Inability to provide informed consent or unwilling to participate
4. Evidence of untreated infection e.g. clostridium difficile
5. Presence of stoma or J pouch
6. Presence of enterocutaneous, abdominal or pelvic fistulae with abscesses or fistulae likely to require surgery during the study period
7. Bowel surgery within 12 weeks prior to screen and/or has surgery planned or deemed likely for IBD during the study period
8. Fixed symptomatic stenosis of small bowel or colon
9. Chronic use of narcotics for chronic pain defined as a daily use of one or more doses of narcotic containing medication
10. Use of oral or intravenous antibiotics within 4 weeks prior to screening
11. Use of tube or enteral feeding, elemental diet, or parenteral alimentation within 2 weeks prior to screening.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | Week 6
  Harvey Bradshaw index < 4 or SCCAI < 3 at week 6

SECONDARY OUTCOMES:
Clinical response | Week 6
  reduction in HBI by 3 or more or SCCAI by 2 or more
Biochemical response - CRP | Week 6
  Change in serum C-reactive protein from baseline
Biochemical response - fecal calprotectin | Week 6
  Change in fecal calprotectin from baseline

OTHER OUTCOMES:
Change in gut microbiome | Week 6 and Week 12
  Change in fecal microbiome pattern assessed using 16sRNA sequencing and shotgun metagenomic sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States